CLINICAL TRIAL: NCT03580902
Title: A Method to Increase Buprenorphine Treatment Capacity
Brief Title: CBT4CBT for Office Based Buprenorphine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CBT4CBT, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41941
Record Dates: First submitted 2018-06-25; First posted 2018-07-10 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Buprenorphine (Active Comparator): Participants assigned to this arm will received buprenorphine treatment consistent with standard practice at the study site. This includes induction by a physician, regular meetings with a physician for medical management, urine monitoring, and prescription of buprenorphine, with access to behavioral support services.
  Interventions: Drug: Buprenorphine/naloxone
- Standard Buprenorphine plus CBT4CBT-Buprenorphine (Experimental): Participants in this condition will receive Standard Buprenorphine as described above, with the addition of access to the CBT4CBT-Buprenorphine program, which is a web-based program that covers basic knowledge about buprenorphine treatment as well as teaches cognitive and behavioral coping skills.
  Interventions: Behavioral: CBT4CBT-Buprenorphine; Drug: Buprenorphine/naloxone

INTERVENTIONS:
Behavioral: CBT4CBT-Buprenorphine — Computerized, user-driven cognitive-behavioral therapy (CBT) web-based program adapted for use in office based buprenorphine treatment
  Arms: Standard Buprenorphine plus CBT4CBT-Buprenorphine
Drug: Buprenorphine/naloxone — Standard outpatient buprenorphine maintenance

SUMMARY:
In this Phase II SBIR/STTR project, our Specific Aim will be to determine if the use of CBT4CBT-Buprenorphine leads to clinically significant improved outcomes and increased retention for buprenorphine maintenance patients in a larger and diverse population of individuals seeking buprenorphine treatment in primary care (N=100).

DETAILED DESCRIPTION:
In this phase, 100 individuals entering buprenorphine maintenance at the primary care clinic (Central Medical Unit, CMU) will be randomized to either (1) standard buprenorphine maintenance in which counseling is offered on site, or (2) standard buprenorphine maintenance with CBT4CBT-Buprenorphine substituting for on-site counseling. This will be a 12-week trial.

ELIGIBILITY:
Inclusion Criteria:

* Meets current Diagnostic Statistical Manual (DSM-5) criteria for opioid use disorder
* Requesting buprenorphine maintenance treatment at Central Medical Unit of the APT Foundation

Exclusion Criteria:

* Unstabilized psychotic disorder
* Currently suicidal or homicidal
* Current cocaine, benzodiazepine, or alcohol use disorder.
* Any history of PCP (phencyclidine) use.
* Pregnant or lactating
* Any other physical or mental condition that would contraindicate office-based buprenorphine maintenance treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Percent of urine toxicology screens that are negative for opioids by group. | 12 weeks
  Percent of urine toxicology screens, collected weekly, that are negative for opioid metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Shi, MD, Principal Investigator — APT Foundation, Inc.
Locations (1):
- Central Medical Unit of the APT Foundation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No